CLINICAL TRIAL: NCT06554353
Title: Cardiopulmonary Exercise Testing and Oscillometry for the Evaluation of Dyspnea
Acronym: COED
Status: Recruiting | Type: Observational
Sponsor: University of Rochester (Other)
Responsible Party: Principal Investigator, Patrick Donohue, Assistant Professor, University of Rochester
Other Study IDs: STUDY00009729
Record Dates: First submitted 2024-08-12; First posted 2024-08-15 (Actual); Last update posted 2025-12-08 (Actual); Status verified 2025-10

CONDITIONS: Breathing, Mouth; Lung Function Decreased; Dyspnea; Shortness of Breath
MeSH Terms: conditions — Mouth Breathing; Respiratory Insufficiency; Dyspnea

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: No

GROUPS / COHORTS (1):
- Subjects with dyspnea referred for Cardiopulmonary Exercise Testing: Subjects with unexplained dyspnea referred for Cardiopulmonary Exercise Testing.
  Interventions: Device: Oscillometer

INTERVENTIONS:
Device: Oscillometer — The tremoFlo C-100 Airwave Oscillometry System is intended to measure respiratory system impedance using the Forced Oscillation Technique (FOT).
  Other Names: THORASYS tremoFlo C-100 Airwave Oscillometry System

SUMMARY:
This study will determine if airway resistance to airflow and pressure, measured by Oscillometry, is associated with abnormal findings on Cardiopulmonary Exercise Testing in subjects who are experiencing shortness of breath.

ELIGIBILITY:
Inclusion Criteria:

* Willingness to perform breathing test
* Must be able to speak and understand English
* Referred for Cardiopulmonary Exercise Testing

Exclusion Criteria:

* Unable to provide consent or perform oscillometry test

Min Age: 18 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: Up to fifty (50) human subjects will be recruited from the following University of Rochester locations: Mary Parkes Center for Asthma, Allergy, and Pulmonary Care, the Pulmonary Clinic at Strong Memorial Hospital, and The Pulmonary Clinic at Highland Hospital.
Sampling Method: Non-Probability Sample
Enrollment: 50 (Estimated)
Dates: Start 2024-10-29 (Actual); Primary Completion 2026-05-01 (Estimated); Study Completion 2026-06-30 (Estimated)

PRIMARY OUTCOMES:
Mean respiratory system resistance and reactance | Single measurement, approximately day 1
  The oscillometer will collect an airway impedance measurement which is made up of multiple variables.

CONTACTS AND LOCATIONS:
Locations (1):
- Highland Hospital, Rochester, New York, United States

IPD SHARING:
Plan to Share IPD: Undecided